CLINICAL TRIAL: NCT00042835
Title: A Phase I Study Of OSI-774 (NSC #718781)-Based Multimodality Therapy For Inoperable Stage III Non Small Cell Lung Cancer
Brief Title: Erlotinib and Radiation Therapy Plus Combination Chemotherapy in Treating Patients With Inoperable Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2012-02478; 11432B; N01CM17102 (NIH); N01CM62201 (NIH); CDR0000069474 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Lung; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Erlotinib Hydrochloride; Radiotherapy; Radiation; Docetaxel; Paclitaxel; Taxes; Carboplatin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Group I (cisplatin, etoposide, erlotinib, and docetaxel) (Experimental): Patients receive cisplatin IV over 2 hours on days 1, 8, 29, and 36; etoposide IV over 1 hour on days 1-5 and 29-33; and oral erlotinib once daily on days 1-49. Patients undergo concurrent radiotherapy 5 days a week for 7 weeks beginning on day 1. Patients receive consolidation therapy comprising docetaxel IV over 1 hour on days 50, 71, and 92. Some patients may also receive oral erlotinib once daily on days 50-112.
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: erlotinib hydrochloride; Radiation: radiation therapy; Drug: docetaxel; Other: laboratory biomarker analysis
- Group II (paclitaxel, carboplatin, and erlotinib (Experimental): Patients receive induction chemotherapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1 and 21. Patients receive consolidation therapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 43, 50, 57, 64, 71, 78, and 85 and oral erlotinib once daily on days 43-91. Patients undergo radiotherapy concurrently with consolidation therapy 5 days a week for 7 weeks beginning on day 43.
  Interventions: Drug: erlotinib hydrochloride; Radiation: radiation therapy; Drug: paclitaxel; Drug: carboplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Group I (cisplatin, etoposide, erlotinib, and docetaxel)
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Group I (cisplatin, etoposide, erlotinib, and docetaxel)
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
  Arms: Group I (cisplatin, etoposide, erlotinib, and docetaxel)
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Group II (paclitaxel, carboplatin, and erlotinib
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Group II (paclitaxel, carboplatin, and erlotinib
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib and radiation therapy with combination chemotherapy may kill more tumor cells. Phase I trial to study the effectiveness of combining erlotinib and radiation therapy with combination chemotherapy in treating patients who have inoperable stage III non-small cell lung cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of erlotinib that can be administered with chest radiotherapy in combination with cisplatin and etoposide or carboplatin and paclitaxel in patients with inoperable stage III non-small cell lung cancer.

II. Determine the dose-limiting toxicity of these regimens in these patients. III. Assess the clinical response (complete response, partial response, progressive disease, or stable disease) in patients treated with these regimens.

IV. Determine levels of tumor epidermal growth factor expression in patients treated with these regimens.

OUTLINE: This is a multicenter, dose-escalation study of erlotinib. Patients are assigned to 1 of 2 treatment groups.

GROUP 1: Patients receive cisplatin IV over 2 hours on days 1, 8, 29, and 36; etoposide IV over 1 hour on days 1-5 and 29-33; and oral erlotinib once daily on days 1-49. Patients undergo concurrent radiotherapy 5 days a week for 7 weeks beginning on day 1. Patients receive consolidation therapy comprising docetaxel IV over 1 hour on days 50, 71, and 92. Some patients may also receive oral erlotinib once daily on days 50-112.

GROUP 2: Patients receive induction chemotherapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1 and 21. Patients receive consolidation therapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 43, 50, 57, 64, 71, 78, and 85 and oral erlotinib once daily on days 43-91. Patients undergo radiotherapy concurrently with consolidation therapy 5 days a week for 7 weeks beginning on day 43.

In both groups, cohorts of 3-6 patients receive escalating doses of erlotinib during concurrent chemoradiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 6 patients experience dose-limiting toxicity. At least 12 patients from each group are treated at the MTD.

Patients are followed at 8 weeks.

PROJECTED ACCRUAL: A total of 24-48 patients (12-24 per treatment group) will be accrued for this study within 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar)
  * Large cell carcinoma (including giant and clear cell carcinomas)
* Stage IIIA (T1 or T2, N2) or IIIB disease not amenable to resection or surgery
* T3, N2 or T4, N0-N2 disease also allowed if based on the closeness to the carina, invasion of the mediastinum, or invasion of the chest wall
* T3, N0-N1 disease allowed provided the disease is not amenable for surgical resection
* No M1 disease
* No disease invasion of a vertebral body

  * Tumors adjacent to a vertebral body allowed provided all gross disease can be encompassed in the radiotherapy boost field and there is no bone invasion
* Contralateral mediastinal disease (N3) allowed if all gross disease can be encompassed in the radiotherapy boost field
* Pleural effusion that is transudative, cytologically negative, and non-bloody allowed if the tumor can be encompassed in a reasonable field of radiotherapy

  * No exudative, bloody, or cytologically malignant effusions
  * Effusions present on CT scans but not on chest x-ray (CXR) and too small for thoracentesis are allowed
* Measurable or evaluable disease

  * Pleural effusions are not considered measurable or evaluable
  * Measurable disease is defined as any mass in 2 perpendicular diameters by CXR, CT scan, or MRI
  * Evaluable disease includes lesions apparent on CXR or CT scan that are:

    * Ill-defined masses associated with post-obstructive changes
    * Mediastinal or hilar adenopathy measurable in only one dimension
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* More than 6 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST and ALT no greater than 1.5 times upper limit of normal (ULN) and alkaline phosphatase normal
* AST and ALT normal and alkaline phosphatase no greater than 2.5 times ULN
* Creatinine normal
* Creatinine clearance at least 50 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of cornea abnormalities (e.g., dry-eye syndrome, Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No gastrointestinal tract disease resulting in the inability to take oral medications
* No required IV alimentation
* No peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergy to compounds of similar chemical or biologic composition to erlotinib or other study agents
* No significant traumatic injury within the past 21 days
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other active malignancy within the past 6 months except non-melanoma skin cancer
* No concurrent colony-stimulating factors (filgrastim [G-CSF] or sargramostim [GM-CSF]) with radiotherapy
* No prior chemotherapy for lung cancer
* See Disease Characteristics
* No prior chest radiotherapy
* See Disease Characteristics
* At least 7 days since prior mediastinoscopy
* More than 3 weeks since prior formal exploratory thoracotomy
* More than 3 weeks since prior major surgery
* No prior surgical procedures affecting absorption
* No prior epidermal growth factor receptor-targeting therapies
* No other concurrent investigational or commercial agents or therapies directed at malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-05; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose at which at least 2 of 6 patients experience dose-limiting toxicity assessed using NCI CTCAE version 3.0 | 7 weeks

SECONDARY OUTCOMES:
Response assessed using RECIST | Up to 8 weeks
Level of EGFR expression | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mauer, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States